CLINICAL TRIAL: NCT02377323
Title: Real-Life Outcomes of Multiple Sclerosis Treatment With Rebif on Employment Status, Quality of Life and Cognition: a Pilot Study
Brief Title: Real-Life Outcomes of Multiple Sclerosis Treatment With Rebif
Acronym: RLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: EMD Serono Canada Inc. (Industry)
Responsible Party: Principal Investigator, Pierre Duquette, MD, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NE156
Record Dates: First submitted 2014-07-31; First posted 2015-03-03 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Patient-reported outcomes; Employment status; Quality of Life; Cognition; Rebif
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with Rebif (Other): Patients treated with Rebif only, for at least two years, and for up to 18 years
  Interventions: Other: MACFIMS; Other: MSQoL-54
- Never treated (Other): Patients never treated with a disease-modifying drug (DMD)
  Interventions: Other: MACFIMS; Other: MSQoL-54

INTERVENTIONS:
Other: MACFIMS — Cognitive evaluation of 50 participants
Other: MSQoL-54 — Quality of life questionnaires

SUMMARY:
The purpose of this study is to determine whether Rebif has an impact on employment status, quality of life and cognition.

DETAILED DESCRIPTION:
With this study the investigator plans to evaluate the impact of Rebif on the Real-Life Outcomes (RLO) of Multiple Sclerosis (MS) patients followed at the Clinic within the last two years, and with a follow-up of up to 18 years.

The investigator will evaluate the employment outcomes with a questionnaire designed to document eventual changes in the employment status and other variables in the work conditions of the study participants.

Furthermore, to evaluate the quality of life (QoL),eligible patients will be asked to complete the Multiple Sclerosis Quality of Life (MSQOL)-54 Instrument, contains 52 items distributed into 12 scales, and two single items. This MS-specific QoL assessment tool uses the Short Form Health Survey (SF-36) as its generic core measure and includes 18 additional items under the following categories: health distress, sexual function, satisfaction with sexual function (one item), overall quality of life, cognitive function, energy, pain, and social function.

A sub-group of patients will be selected to come to the clinic to undergo the cognitive portion of the study, using the well-known and validated battery of tests named Minimal Assessment of Cognitive Function in MS (MACFIMS battery).

Socio-demographic data on education level, marital and family life will also be collected. All questionnaires (including the MSQoL-54) will be available by means of an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CIS or definite MS (RRMS or SPMS);
* Patients seen at our Clinic within the last 2 years;
* Patients untreated, or treated with either low dose or high dose Rebif for at least two years;
* Patients between 18 to 60 years old at time of treatment initiation;
* EDSS ≤ 5.5 at treatment initiation;
* Patients able to read and write in French.

Exclusion Criteria:

* Patients diagnosed with primary progressive MS;
* Patients treated with other DMD, other than Rebif;
* Co-existence of other diseases that could influence outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Employment status | baseline
  The primary endpoint is the proportion of patients in each group belonging in the employment categories listed below:
  1. Never worked
  2. Work status unchanged
  3. Work status changed: Not due to MS / Due to MS
  Sub-groups:
  1. Full employment with accommodations
  2. Part-time employment
  3. Complete invalidity
  4. Patient retired

SECONDARY OUTCOMES:
Quality of life | Baseline
  The MSQoL-54 scores of the Rebif treated patient group compared to the never treated patient group.
Cognitive function | Baseline
  The comparison of the score of each patient group using the MACFIMS cognitive function tests.

OTHER OUTCOMES:
Clinical variables - Composite measure | baseline
  The comparison of the clinical variables such as the Kurtzke Expanded Disability Status Scale (EDSS), relapse-rate, MS course and, when available, magnetic resonance imaging (MRI) of each patient group.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Duquette, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- CHUM, Montreal, Quebec, Canada

REFERENCES:
- [Background] Trojano M, Pellegrini F, Paolicelli D, Fuiani A, Zimatore GB, Tortorella C, Simone IL, Patti F, Ghezzi A, Zipoli V, Rossi P, Pozzilli C, Salemi G, Lugaresi A, Bergamaschi R, Millefiorini E, Clerico M, Lus G, Vianello M, Avolio C, Cavalla P, Lepore V, Livrea P, Comi G, Amato MP; Italian Multiple Sclerosis Database Network (MSDN) Group. Real-life impact of early interferon beta therapy in relapsing multiple sclerosis. Ann Neurol. 2009 Oct;66(4):513-20. doi: 10.1002/ana.21757. PMID 19847899
- [Background] Glanz BI, Degano IR, Rintell DJ, Chitnis T, Weiner HL, Healy BC. Work productivity in relapsing multiple sclerosis: associations with disability, depression, fatigue, anxiety, cognition, and health-related quality of life. Value Health. 2012 Dec;15(8):1029-35. doi: 10.1016/j.jval.2012.07.010. Epub 2012 Oct 25. PMID 23244804
- [Background] Krokavcova M, Nagyova I, Van Dijk JP, Rosenberger J, Gavelova M, Middel B, Szilasiova J, Gdovinova Z, Groothoff JW. Self-rated health and employment status in patients with multiple sclerosis. Disabil Rehabil. 2010;32(21):1742-8. doi: 10.3109/09638281003734334. PMID 20350069
- [Background] Roessler RT, Rumrill PD Jr. Multiple sclerosis and employment barriers: a systemic perspective on diagnosis and intervention. Work. 2003;21(1):17-23. PMID 12897387
- [Background] Beatty WW, Hames KA, Blanco CR, et al. Demographic, clinical and cognitive characteristics of multiple sclerosis patients who continue to work. J Neurol Rehab 1995; 9:167-73.
- [Background] Simmons RD, Tribe KL, McDonald EA. Living with multiple sclerosis: longitudinal changes in employment and the importance of symptom management. J Neurol. 2010 Jun;257(6):926-36. doi: 10.1007/s00415-009-5441-7. Epub 2010 Jan 19. PMID 20084515
- [Background] Larocca N, Kalb R, Scheinberg L, Kendall P. Factors associated with unemployment of patients with multiple sclerosis. J Chronic Dis. 1985;38(2):203-10. doi: 10.1016/0021-9681(85)90093-1. PMID 3156140
- [Background] Smith MM, Arnett PA. Factors related to employment status changes in individuals with multiple sclerosis. Mult Scler. 2005 Oct;11(5):602-9. doi: 10.1191/1352458505ms1204oa. PMID 16193900
- [Background] Verdier-Taillefer MH, Sazdovitch V, Borgel F, Cesaro P, Kurtz A, Millet MF, Roullet E, Marteau R. Occupational environment as risk factor for unemployment in multiple sclerosis. Acta Neurol Scand. 1995 Jul;92(1):59-62. doi: 10.1111/j.1600-0404.1995.tb00467.x. PMID 7572062
- [Background] Glad SB, Nyland H, Aarseth JH, Riise T, Myhr KM. How long can you keep working with benign multiple sclerosis? J Neurol Neurosurg Psychiatry. 2011 Jan;82(1):78-82. doi: 10.1136/jnnp.2010.210732. Epub 2010 Aug 27. PMID 20802029
- [Background] Rao SM, Leo GJ, Ellington L, Nauertz T, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. II. Impact on employment and social functioning. Neurology. 1991 May;41(5):692-6. doi: 10.1212/wnl.41.5.692. PMID 1823781
- [Background] Benito-Leon J, Morales JM, Rivera-Navarro J, Mitchell A. A review about the impact of multiple sclerosis on health-related quality of life. Disabil Rehabil. 2003 Dec 2;25(23):1291-303. doi: 10.1080/09638280310001608591. PMID 14617435
- [Background] Rudick RA, Miller D, Clough JD, Gragg LA, Farmer RG. Quality of life in multiple sclerosis. Comparison with inflammatory bowel disease and rheumatoid arthritis. Arch Neurol. 1992 Dec;49(12):1237-42. doi: 10.1001/archneur.1992.00530360035014. PMID 1449401
- [Background] Kobelt G, Berg J, Lindgren P, Kerrigan J, Russell N, Nixon R. Costs and quality of life of multiple sclerosis in the United Kingdom. Eur J Health Econ. 2006 Sep;7 Suppl 2:S96-104. doi: 10.1007/s10198-006-0380-z. PMID 17310341
- [Background] Solari A. Role of health-related quality of life measures in the routine care of people with multiple sclerosis. Health Qual Life Outcomes. 2005 Mar 18;3:16. doi: 10.1186/1477-7525-3-16. PMID 15777478
- [Background] Amato MP, Zipoli V, Portaccio E. Multiple sclerosis-related cognitive changes: a review of cross-sectional and longitudinal studies. J Neurol Sci. 2006 Jun 15;245(1-2):41-6. doi: 10.1016/j.jns.2005.08.019. Epub 2006 Apr 27. PMID 16643953
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Background] Amato MP, Ponziani G, Pracucci G, Bracco L, Siracusa G, Amaducci L. Cognitive impairment in early-onset multiple sclerosis. Pattern, predictors, and impact on everyday life in a 4-year follow-up. Arch Neurol. 1995 Feb;52(2):168-72. doi: 10.1001/archneur.1995.00540260072019. PMID 7848126
- [Background] Kujala P, Portin R, Ruutiainen J. The progress of cognitive decline in multiple sclerosis. A controlled 3-year follow-up. Brain. 1997 Feb;120 ( Pt 2):289-97. doi: 10.1093/brain/120.2.289. PMID 9117376
- [Background] Jennekens-Schinkel A, Laboyrie PM, Lanser JB, van der Velde EA. Cognition in patients with multiple sclerosis After four years. J Neurol Sci. 1990 Nov;99(2-3):229-47. doi: 10.1016/0022-510x(90)90158-j. PMID 2086726
- [Background] Amato MP, Ponziani G, Siracusa G, Sorbi S. Cognitive dysfunction in early-onset multiple sclerosis: a reappraisal after 10 years. Arch Neurol. 2001 Oct;58(10):1602-6. doi: 10.1001/archneur.58.10.1602. PMID 11594918
- [Background] Benedict RH, Cookfair D, Gavett R, Gunther M, Munschauer F, Garg N, Weinstock-Guttman B. Validity of the minimal assessment of cognitive function in multiple sclerosis (MACFIMS). J Int Neuropsychol Soc. 2006 Jul;12(4):549-58. doi: 10.1017/s1355617706060723. PMID 16981607
- [Background] Fischer JS, LaRocca NG, Miller DM, Ritvo PG, Andrews H, Paty D. Recent developments in the assessment of quality of life in multiple sclerosis (MS). Mult Scler. 1999 Aug;5(4):251-9. doi: 10.1177/135245859900500410. PMID 10467384
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530